CLINICAL TRIAL: NCT02790281
Title: A Study to Investigate Interleukin-6 (IL-6) and IL-6/Soluble IL-6 Receptor (sIL-6R) Complex Levels in Subjects With Active Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 07031-01
Record Dates: First submitted 2016-05-18; First posted 2016-06-03 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Blood sampling — Blood sample collected at a single visit

SUMMARY:
The purpose of this study is to measure IL-6 and IL-6/sIL-6R complex levels in subjects with active moderate to severe ulcerative colitis or Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with active moderate to severe ulcerative colitis (*partial Mayo ≥ 5) or Crohn's disease (Harvey & Bradshaw ≥ 8) *partial Mayo: 9-point scale that excludes the endoscopic components of the Mayo score

Exclusion Criteria:

* Presence of another inflammatory disease, except for mild cutaneous psoriasis
* Concomitant gastrointestinal infection or otherwise serious infection including Crohn's disease infectious complication
* Treatment with Infliximab, Adalimumab, Certolizumab Pegol or other immune-modulating biologics within 8 weeks prior to the visit
* Having a known or suspected gastrointestinal or otherwise serious infection within 8 weeks prior to the visit
* Concomitant diagnosed or suspected malignant disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men and women seeking medical support due to present, active moderate to severe ulcerative colitis or Crohn's disease (newly diagnosed or during disease relapse).
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (2):
- Herlev hospital (there may be other sites in this country), Herlev, Denmark
- Skane University Hospital (there may be other sites in this country), Lund, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from amongst the subjects seeking medical support due to present, active moderate to severe ulcerative colitis or Crohn's disease (newly diagnosed or during disease relapse) at four sites in two countries (Denmark and Sweden) between 10 Dec 2014 to 20 Aug 2015.
Groups:
- Overall Study: Subjects included were diagnosed with active moderate to severe ulcerative colitis or Crohn's disease and C-reactive protein (CRP) >5 mg/L.
Period: Overall Study
Arm/Group | Overall Study
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set, consisted of all eligible subjects with CRP >5 mg/L.
Arm/Group | Overall Study
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (16.41)
Gender [Count of Participants; unit: Participants]
  Female | 16
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Exploratory: Levels of IL-6/sIL-6R Complex
Description: Blood sample was taken for analysis of levels of IL-6/sIL6-R complex.
Time Frame: At Day 1
Population: All eligible subjects with CRP >5 mg/L.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Overall Study
Number analyzed (Participants) | 33
pg/mL | NA [NA to NA] — Levels of IL-6/sIL6-R complex were below level of detection.

2. Primary Outcome: Exploratory: Levels of IL-6
Description: Blood sample was taken for analysis of levels of IL-6.
Time Frame: At Day 1
Population: All eligible subjects with CRP >5 mg/L
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Overall Study
Number analyzed (Participants) | 33
pg/mL | NA [NA to NA] — Levels of IL-6 were below level of detection.

3. Primary Outcome: Exploratory: Levels of C-reactive Protein (CRP)
Description: Blood sample was taken for analysis of levels of CRP.
Time Frame: At Day 1
Population: All eligible subjects with CRP >5 mg/L
Measure: Median (Full Range); unit: mg/L
Arm/Group | Overall Study
Number analyzed (Participants) | 33
mg/L | NA [NA to NA] — Levels of CRP were below level of detection.

ADVERSE EVENTS:
Time Frame: No data for adverse event was collected in this study as no investigational medicinal product was administered to the subjects.
Description: Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Manuscripts or abstracts will be prepared in collaboration between Ferring and the Investigators.